CLINICAL TRIAL: NCT06478459
Title: A Single-center, Single-arm, Open-label, Dose-escalation Clinical Study to Evaluate the Safety and Anti-tumor Efficacy of Intratumoral NKG2D CAR-NK Cell Injection Guided by EUS in the Treatment of Locally Advanced Pancreatic Cancer.
Brief Title: Endoscopic Ultrasound (EUS) Intratumoral Injection of CAR-NK Cells in the Treatment of Advanced Pancreatic Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-C1/22A1-08
Record Dates: First submitted 2024-06-09; First posted 2024-06-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-06

CONDITIONS: Pancreatic Cancer Non-resectable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAR-NK：intratumoral injection combined with intravenous infusion (Experimental)
  Interventions: Biological: CAR-NK

INTERVENTIONS:
Biological: CAR-NK — Endoscopic ultrasound-guided intratumoral CAR-NK injection once at day 0, combined with intravenous CAR-NK infusion twice at day 4 and 5

SUMMARY:
This is a single-center, single-arm, open-label, dose-escalation clinical study to evaluate the safety and anti-tumor efficacy of intratumoral NKG2D CAR-NK cell injection guided by endoscopic ultrasound in the treatment of locally advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. 18~75 years old (including boundary value), both male and female.
2. Histologically or cytologically confirmed pancreatic ductal adenocarcinoma or IPMN carcinogenesis.
3. Recurrent or unresectable locally advanced pancreatic cancer. Patients with technically resectable tumors but are considered as unable to undergo surgical treatment due to medical comorbidities or the patient's refusal of surgery are also eligible for enrollment.
4. ECOG PS score of 0-1.
5. At least 3 months of life expectancy at screening, as judged by the investigator.
6. Subject has adequate organ and bone marrow function. Laboratory screening results should be within the stable range described below, and there should be no ongoing supportive care ("jaundice relieve" therapy such as PTCD, ENBD, or bile duct stenting is allowed when pancreatic cancer invades the common bile duct). a) Blood biochemistry: serum creatinine ≤ 1.5×ULN, serum total bilirubin ≤ 2.0×ULN, and serum liver aminotransferase ≤ 3 ×ULN b) Blood tests: neutrophil count ≥ 1.5×109/L, platelet count ≥ 60×109/L, hemoglobin ≥ 8.0g/dL, lymphocyte count ≥ 0.4×109/L;
7. Childbearing status: not pregnant and, if of childbearing potential, willing to use effective contraception from the time of signing the informed consent form until 6 months after the last cell infusion (women of childbearing potential include premenopausal women and women within 2 years of postmenopausal time).
8. Subjects must sign a written informed consent form.
9. Subjects must be voluntary and able to comply with the scheduled treatment regimen, laboratory tests, follow-up, and other study requirements.

Exclusion Criteria:

1. Pregnant and lactating females.
2. Received any anti-tumor therapy (including but not limited to radiotherapy, chemotherapy, or immunotherapy) for pancreatic cancer within 28 days prior to enrollment.
3. In the opinion of the investigator, the EUS technique poses undue risks to the subject, including but not limited to: - Previous EUS-FNA was technically deemed too difficult to perform; - Imaging showing multiple collateral vessels around or near the target tumor within the pancreas; - Presence of varicose veins near the target tumor. - If any of the above risk profiles become apparent after subject screening and/or enrollment, consideration should be given to withdrawal from the study prior to treatment.
4. History of malignancy within 5 years, with the exception of basal cell carcinoma of the skin and carcinoma in situ of the cervix.
5. Any other health condition by the judgment of the investigator would preclude participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-09 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | within 28 days after NKG2D CAR-NK treatment
  Determine the optimal agent for NKG2D CAR-NK at maximum tolerated dose
Dose limiting toxicity | From enrollment of the first subject to completion of follow-up of the last subject（up to 2 years））
  Describe the adverse events of limiting further increases in the dose of NKG2D CAR-NK

SECONDARY OUTCOMES:
Effectiveness evaluation | At weeks 4，8 and months 3，6，9，12，16，20 and 24 after treatment
  Objective Response Rate (ORR) According to Response Evaluation Criteria In Solid Tumors Version 1.1
Cell continued survival time in vivo | At weeks 4，8 and months 3，6，9，12，16，20 and 24 after treatment
  Detect the copy number of NKG2D CAR DNA in peripheral blood at each visit point after the end of the infusion, until any 2 consecutive test results were negative

CONTACTS AND LOCATIONS:
Locations (1):
- the first affiliated hospital of Zhejiang University，school of medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No